

Faculty of Applied Science



#### For the Research Project:

### Promoting Health Equity for Indigenous and non-Indigenous People in Emergency Departments

## **Consent Form Patient Survey**

Principal Investigators: Colleen Varcoe (UBC), Annette J. Browne (UBC), Victoria Bungay (UBC), David W. Byres (Providence Health Care), Roberta Price (UBC)

Co-Investigators: Agnes Black (Providence Health Care), Amélie Blanchet Garneau (UBC), Gary Scott Comber (Dalhousie University), Alison Gerlach (UBC), Emily Jenkins (UBC), Bindy Kang (UBC), Lorraine Prysunka (Fraser Health), Heather Smith (UHNBC), Erin Wilson (University of Northern British Columbia)

Funded by: Canadian Institutes of Health Research (CIHR)

#### Invitation

You are being invited to participate in a research study. The goal of the study is to help improve care for all people who come to this Emergency Department (ED).

We invite you to participate in this study by completing a survey with us. The survey asks your opinions about the care you receive during this ED visit. We plan to survey about 4500 patients at three emergency departments over the next few years.

To participate, you must be an adult (age 19 or older) or emancipated minor receiving care at this **Emergency Department.** 

#### What participating means:

If you agree to participate, a researcher will sit with you to collect your answers on a tablet. There are two parts to the survey. The first part asks some general questions about you (for example, about your overall health and your gender, culture/ethnicity, etc.) and can be completed at any time during your visit to the ED. The second part asks your opinions about the health care provided to you (for example, were you treated with courtesy and respect by doctors and nurses), and will be completed at the end of your ED visit. You will have the option to complete the second part before you leave the hospital or within 2 – 5 days by phone or at a nearby location.













#### **School of Nursing** Faculty of Applied Science

The survey has two sections, and each section should take about 10 to 15 minutes to complete. To thank you for your time, you will be paid \$10 for each section of the survey (up to \$20). If you choose to complete the second part in-person after leaving the Emergency Department, we can also pay for any childcare, dependent care or travel costs. You may keep this money even if you stop participating in the study.

We will not delay or interfere with your care in any way. If you are in need of immediate medical attention, we will not talk with you until after you have received that attention.

Taking part in this study is your choice. You can stop the survey at any time and can refuse to answer or skip over specific questions. Whether you choose to participate or not will not affect how quickly you are seen. It will not affect your care or your ability to get the care you need.

#### **Privacy and Confidentiality:**

Information collected is strictly confidential and will not affect your care in any way.

Your name will not be attached to the information collected in this study. Instead, a number code will be given to each person in the study.

Staff at this hospital will not know if you choose to participate in the survey or not. They will not be able to see, read, or hear anything you say to a researcher in a way that will identify you.

Your name will never be used in any reports of this research. What you tell us will be used for final reports, articles in magazines and professional journals, and public talks. The results from this study may be used by researchers in future projects. Please let the researchers know if you would like a report of what we learn.

All information will be stored securely in a locked cabinet or password-protected computer in a research office at University of British Columbia. Your name and contact information will be kept separately from your survey responses. All research materials will be stored for at least 5 years after the work is published or presented. After that time, digital and paper records may be securely destroyed.

During the survey, you and a researcher will enter your responses on a tablet using the UBC Survey Tool, which is a Canadian-hosted survey solution complying with the BC Freedom of Information and Protection of Privacy Act (FIPPA).

Your confidentiality will be respected. However, research records identifying you may be inspected in the presence of the Investigator or her designate by representatives of the Providence Health Research Ethics Board, the Fraser Health Research Ethics Board, or the Northern Health Research Review Committee for the purpose of monitoring the research. No information or records that disclose your identity will be published without your consent, nor will any information or records that disclose your identity be removed or released without your consent unless required by law.













## **School of Nursing**

Faculty of Applied Science

Even if you decide to stop participating, the information you have provided will be kept and may be used in this study, unless you specifically request otherwise.

#### **Potential Risks and Benefits:**

There are no risks to your health from taking part in this study. Other risks are small. Talking about your health and the health care you receive may be upsetting. If you become upset, support will be provided. If you wish, we will give you information to help you get counselling or other support services.

The survey will give you a chance to share your thoughts and experiences about your health and the care given to you at this Emergency Department. What you share with us may help health care providers, staff, and policy makers to improve the quality of care. You will not directly benefit from participation in this study.

## Questions about this study:

If you have any questions about the study, please call Phoebe Long, Research Manager, at 604-822-3183 (1-844-822-3183 toll-free), or Colleen Varcoe, Professor, University of British Columbia, at 604-827-3121.

If you have any concerns or complaints about your rights as a research participant and/or your experiences while participating in this study, please contact:

- Research Participant Complaint Line in the UBC Office of Research Ethics at 604-822-8598 or if long distance e-mail RSIL@ors.ubc.ca or call toll free 1-877-822-8598;
- Fraser Health Research Ethics Board co-Chair by calling 604-587-4681; or
- Northern Health Research Review Committee by calling 250-649-7598 or by email to researchcommittee@northernhealth.ca.

This letter is for you to keep.













Faculty of Applied Science

## For the Research Project:

# Promoting Health Equity for Indigenous and non-Indigenous People in Emergency Departments

| Consent | | |
|---|---|---|
| Your participation in this survey is completely voluntary. | | |
| If you decide to participate in the study and then change your mind, you are free to withdraw at any time with no consequence. | | |
| By signing this consent form you agree<br>any of your legal rights. You have recei | | _ |
| Signature of Participant | Printed Name | Date |
| Signature of Principal Investigator or designate | Printed Name | Date |









